CLINICAL TRIAL: NCT02984150
Title: Effect of Intragastric Administration of Fatty Acids on Generalized Reward Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S55265
Record Dates: First submitted 2016-10-24; First posted 2016-12-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — lauric acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- fatty acid (Experimental): the nutrient that can be widely found in daily food.
  Interventions: Dietary Supplement: dodecanoic acid
- saline (Sham Comparator): saline
  Interventions: Dietary Supplement: saline

INTERVENTIONS:
Dietary Supplement: dodecanoic acid
  Other Names: Lauric acid
  Arms: fatty acid
Dietary Supplement: saline
  Arms: saline

SUMMARY:
This study aim to investigate the influence of intragastrically infused fatty acid on the generalization of responses to reward within the food domain and between financial and sexual domains.

DETAILED DESCRIPTION:
Earlier research at the Faculty of Economics and Business (FEB) has demonstrated generalization of reward sensitivity after sensory stimulation in a different domain. As increased sensory stimulation in the sexual domain (Van den Bergh et al. 2008) or the power domain (Briers et al. 2007), the preference for immediate small financial reward increased deferred pay. Hongda, DeWitte & Warlop (2008) were able to neutralize this effect by domain-specific financial satiation. In this research, The investigators investigate the possible influence of (subliminal) intragastric administration of fatty acids in reward sensitivity in the power domain, and whether this effect generalizes to financial and sexual domain. Previous research at the Translational Research Center for Gastrointestinal Disorders (TARGID) showed that such administration can neutralize the effects of mood-priming (Van Oudenhove et al., 2011). This study aims to examine the implications of those findings in the motivational domain.

60 healthy heterosexual men come to the lab twice, once for the fatty acid condition, once for the control condition (counterbalanced, and randomly assigned to sequence condition). In each session the same dv's are measured (first three tasks counterbalanced, progressive ratio task always at the end). At the end of the second session, participants also compete a series of interindividual difference measures (scales).

This research forms the start of a collaboration between TARGID and the Center for Research in Marketing and Consumer Science at KU Leuven Faculty of Business and Economics. The current paradigm is largely based on an earlier study by Prof. Dr. Lukas Van Oudenhove showing the effect of intragastric administration of an identical fatty acid solution tested for mood regulation (Van Oudenhove et al., 2011). The procedure performed in this study, which is placing a thin nasogastric tube is frequently used in the TARGID research and other research and is absolutely proven to be safe, with no mention of any adverse reactions during numerous previous studies. Similar studies by our research group had already been approved by the Medical Ethics Committee, and as always sees Prof. Tack ensure that the study conducted by researchers who have received adequate training and have acquired sufficient experience in this specific procedure before the start of the study. The procedure can be carried out in healthy volunteers in a perfectly safe manner.

ELIGIBILITY:
Inclusion Criteria:

* Men, self-reporting as heterosexual
* Age: Adults (+ 17yr)
* 19 ≤ BMI ≤ 27

Exclusion Criteria:

* Participants must be in good health, both mental and physical. People with one or more of the following self-reported items applicable, are excluded:

  1. History of or current presence of:
* Psychiatric disorders (among others, anxiety disorders, somatoform disorders, eating disorders, depression, addiction-related disorders, and the like)
* Abdominal / Thoracic Surgery (excl appendectomy or cholecystectomy)
* Neurological, endocrine or gastrointestinal-related disorders
* Other serious medical conditions.

  2. Present the presence of:
* Pain Symptoms
* Use of medication that affects the function of the gastrointestinal tract and / or the nervous system; psychotropic drugs or pain killers
* A recent accident or an operation which one has not yet fully recovered.

If it is positive answer to any of these criteria, participation will not be possible. These criteria are questioned in advance so that participants do not get unnecessarily turn up.

Min Age: 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
progressive ratio task | 10min
  Participants click the screens to get candies. The number of clicks will be used as a measurement of eating behavior.
estimation task | 10min
  Participants rate the attractiveness of 20 rewarding food pictures, 20 female face pictures on a 1-7 point scale.

SECONDARY OUTCOMES:
VAS | 10min
  participants rate their appetite related pictures on 100-point scale

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, campus Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Briers, B., Pandelaere, M. & Warlop, L. (2007). Adding exchange to charity: A reference price explanation. Journal of Economic Psychology, 28, 15-30. doi: 10.1016/j.joep.2005.12.001.
- [Background] Lassman DJ, McKie S, Gregory LJ, Lal S, D'Amato M, Steele I, Varro A, Dockray GJ, Williams SC, Thompson DG. Defining the role of cholecystokinin in the lipid-induced human brain activation matrix. Gastroenterology. 2010 Apr;138(4):1514-24. doi: 10.1053/j.gastro.2009.12.060. Epub 2010 Jan 18. PMID 20080096
- [Background] Van den Bergh, B., Dewitte, S. & Warlop, L. (2008). Bikinis instigate generalized impatience in intertemporal choice. Journal of Consumer Behavior, 35, 85-97. doi: 10.1086/525505
- [Background] Van Oudenhove L, McKie S, Lassman D, Uddin B, Paine P, Coen S, Gregory L, Tack J, Aziz Q. Fatty acid-induced gut-brain signaling attenuates neural and behavioral effects of sad emotion in humans. J Clin Invest. 2011 Aug;121(8):3094-9. doi: 10.1172/JCI46380. Epub 2011 Jul 25. PMID 21785220